CLINICAL TRIAL: NCT03617406
Title: Volume Challenge Added to Dobutamine Stress Echocardiography in the Diagnosis of Severe Low-Flow, Low-Gradient Aortic Stenosis
Brief Title: Volume Challenge Added to DSE in the Diagnosis of Severe LFLGAS
Acronym: FLOW-AS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3635
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Aortic Valve Stenosis
Keywords: Low - flow; Low - gradient; Low - dose dobutamine; Volume challenge; Echocardiography
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm Volume Challenge (Other): A standard LDDSE will be performed. The stroke volume (SV) will be recorded. The addition of VC with the passive leg raise method at peak dobutamine dose will be performed. A TEE with low dose dobutamine and a bolus of normal saline will be performed as a validation method.
  Interventions: Diagnostic Test: Volume Challenge

INTERVENTIONS:
Diagnostic Test: Volume Challenge — Addition volume challenge with passive leg raising method in LDDSE as well as administration of normal saline and dobutamine during TEE

SUMMARY:
The aim of this study is to test the diagnostic added value of Volume Challenge (VC) to low-dose dobutamine stress echocardiography (LDDSE) in patients with a low-flow, low-gradient aortic stenosis (LFLGAS). This study will assess if LDDSE plus VC allows to increase the proportion of patients in whom a true severe AS can be differentiated from a pseudo severe AS.

DETAILED DESCRIPTION:
The design of the study is a monocentric prospective non-randomized pilot clinical trial. A standard LDDSE will be performed. The stroke volume (SV) will be recorded. The addition of VC with the passive leg raise method at peak dobutamine dose will be performed. A transesophageal echocardiography (TEE) with low dose dobutamine and a bolus of normal saline will be performed as a validation method to measure AVA with the planimetry method. The SV will be recorded. Proportion of patient receiving the diagnosis of true severe AS defined as a combination of AVA <1.0 cm2 and ∆SV ≥ 20% will be compared between standard LDDSE and LDDSE with addition of VC. Calculating sensitivity, specificity, performing ROC curve analysis and calculating the Youden-index, the accuracy of the test method (LDDSE plus passive leg raising) for the detection of truly severe AS in comparison with the reference method (TEE) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Written informed consent
* Patients with LFLGAS (mean Gradient: < 40 mmHg, AVA ≤ 1.0 cm2 (by continuity equation using LVOT diameter) SVI ≤ 35 ml/m2), by rest TTE

Exclusion Criteria:

* Hypersensitivity to dobutamine or midazolam
* Lack of safe contraception defined as: Female participants of childbearing potential not using and not willing to continue contraception for study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.,
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Previous enrolment into the current study,

ADDITIONAL SPECIFIC EXCLUSION CRITERIA REGARDING STRESS ECHOCARDIOGRAPHY:

* Systolic left ventricular ejection fraction (LVEF) < 20%
* More than mild aortic regurgitation
* Mitral valve disease, defined by mitral valve area < 2.0 cm2 or more than mild mitral regurgitation
* Unstable angina
* Acute pulmonary oedema
* Signs of relevant left ventricular heart failure defined as crackles more than one fourth of lung field on auscultation
* Signs of relevant right ventricular heart failure defined as central venous pressure (CVP) > 15 mmHg estimated with dilatation and collapsibility of vena cava inferior (VCI)
* Severe pulmonary, renal or hepatic disease

ADDITIONAL SPECIFIC EXCLUSION CRITERIA REGARDING TRANSESOPHAGEAL ECHOCARDIOGRAPHY:

* Oesophageal varices
* History of bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of true severe AS | Measures taken during echocardiograph a few minutes after administration of VC
  Proportion of patients receiving the diagnosis of true severe AS defined as a combination of AVA <1.0 cm2 and ∆SV ≥ 20% will be compared between standard LDDSE and LDDSE with addition of VC

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD, Principal Investigator — University Clinic for Cardiology, Inselspital, Bern; Stefano de Marchi, MD, Study Chair — University Clinic for Cardiology, Inselspital, Bern
Locations (1):
- Bern University hospital, Bern, Switzerland